CLINICAL TRIAL: NCT05932030
Title: Assessment of Knowledge and Perceptions of Artificial Intelligence in Solid Organ Transplantation
Acronym: TransplantIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-A00950-45
Record Dates: First submitted 2023-05-16; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Solid Organ Transplantation; Artificial Intelligence
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients and health professionals (Other): The intervention is a survey administered to patients and health professional. The two questionnaires are identical, with only the socio-demographic section differing. The questionnaire is composed of closed questions, scale scores and short-answer questions.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Submission of a survey to solid organ transplant patients and health professionals working in transplantation to assess their knowledge and perception of the use of artificial intelligence in transplantation

SUMMARY:
The increasing abundance of clinical, genetic, radiological, and metabolic data in transplantation has led to a growing interest in applying artificial intelligence (AI) tools to optimize immunosuppression and overall patient management.

However, the majority of these applications exist only in the preclinical state and the field of artificial intelligence remains unknown to the general public. In view of the potential applications of AI and the growing research interest in this topic, it is essential to assess the knowledge and perceptions of those directly involved in solid organ transplantation.

Primary Objective: To assess the knowledge and perceptions of solid organ transplant patients and healthcare professionals working in the field of solid organ transplantation

Primary endpoint:

* Analysis of verbatim and closed-ended questionnaire data
* Comparison of the averages obtained by the subgroups of patients and health professionals and analysis of the verbatim by grouping them by themes

DETAILED DESCRIPTION:
Solid organ transplantation is the treatment of last resort for end-stage organ disease. In France, 51860 patients receive transplants, and the number of candidates awaiting transplantation has doubled in 10 years. At the same time as considerable progress has been made in recent decades, new challenges have emerged. The growing disparity between demand and supply of organs calls for optimal selection and matching of patients and donors. Improving long-term graft and patient survival requires data-driven diagnosis and management of post-transplant complications. The increasing abundance of clinical, genetic, radiological and metabolic data in transplantation has led to growing interest in applying artificial intelligence (AI) tools to optimize immunosuppression and overall patient management.

However, the majority of these applications are still in the pre-clinical stage, and the field of artificial intelligence remains largely unknown to the general public. In view of the potential applications of AI and the growing research interest in the subject, it is essential to assess the knowledge and perceptions of those directly involved in solid organ transplantation.

This is a prospective, observational, multicenter study. The questionnaire will be submitted face-to-face to healthcare professionals working in solid organ transplantation and solid organ transplant patients at Grenoble Alpes University Hospital. It will be put online on the LimeSurvey platform and offered to healthcare professionals at France's various transplant centers via the federations of each organ specialty, as well as to all organ transplant patients in France via patient associations.

The data included will be collected from paper questionnaires and online on the LimeSurvey platform. They will be stored on a secure server at the TIMC research laboratory department. Data will be anonymized for inclusion in the database. An identifier will be assigned to each volunteer at the time of inclusion.

Categorical data will be reported as frequency, percentage, and continuous data as mean and standard deviation or median and interquartile range if they do not follow a normal distribution. The normality of quantitative variables will be tested by graphical verification.

Continuous variables will be compared using a Student's t test if the conditions of application are valid (or Mann-Whitney if applicable). Categorical variables will be compared using a Chi2 test (or Fisher's test if validity conditions are not met).

We consider p values <0.05 to be significant. Statistical analysis will be carried out using RStudio software (version 4.2.1).

ELIGIBILITY:
Inclusion Criteria:

* age greater than or equal to 18 years
* solid organ transplant patients or health professionals working in transplantation
* no opposition to the study

Exclusion Criteria:

* subject under guardianship or deprived of liberty
* hematopoietic stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6750 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge and perceptions evaluation of solid organ transplant patients and healthcare professionals working with solid organ transplantation | 15 minutes
  Analysis of the verbatim by theme and comparison of the averages of closed questions or scale questions of the questionnaire obtained by the subgroups of patients and health professionals. For scale question studying the knowledge of AI the score goes from 0 to 10 with 0 for no knowledge and 10 for perfect knowledge. A verbatim is the complete reproduction of the words spoken by the interviewee. Verbatim will be grouped by response group and compared.

SECONDARY OUTCOMES:
Level of knowledge comparison between different healthcare professionals on artificial intelligence | 15 minutes
  Comparison of the averages obtained by the different types of health professionals. The average is calculated from the results obtained for the closed questions and the knowledge level score (ranging from 0 to 10, 0 for no knowledge and 10 for perfect knowledge) in the questionnaire.
Perceptions comparison between different healthcare professionals on artificial intelligence | 15 minutes
  Analysis of the verbatim by grouping them by theme. A verbatim is the complete reproduction of the words spoken by the interviewee. Verbatim will be grouped by response group and compared.
Comparison of level of artificial intelligence knowledge of patients based on the transplanted organ | 15 minutes
  Comparison of the averages obtained by patients by transplanted organ. The average is calculated from the results obtained for the closed questions and the knowledge level score (ranging from 0 to 10, 0 for no knowledge and 10 for perfect knowledge) in the questionnaire.
Comparison of the perception on artificial intelligence of patients according to the transplanted organ | 15 minutes
  Analysis of the verbatim by grouping them by theme. A verbatim is the complete reproduction of the words spoken by the interviewee. Verbatim will be grouped by response group and compared.
Comparison of the average level of knowledge about artificial intelligence of healthcare professionals and patients. | 15 minutes
  Comparison of overall averages between patients and health professionals. The average is calculated from the results obtained for the closed questions and the knowledge level score (ranging from 0 to 10, 0 for no knowledge and 10 for perfect knowledge) in the questionnaire.
Comparison of the levels of perception of artificial intelligence among healthcare professionals and patients | 15 minutes
  Analysis of the verbatim by grouping them by theme. A verbatim is the complete reproduction of the words spoken by the interviewee. Verbatim will be grouped by response group and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Pierrick Bedouch, Pr, Principal Investigator — University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: No